CLINICAL TRIAL: NCT04958395
Title: Evaluation of the Hemodynamic Significance of Myocardial Bridge by Coronary Blood Fractional Flow Reserve
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014188
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2014-11

CONDITIONS: Myocardial Bridge
MeSH Terms: conditions — Myocardial Bridging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myocardial bridge: Measure FFR and d-FFR
  Interventions: Diagnostic Test: FFR and d-FFR

INTERVENTIONS:
Diagnostic Test: FFR and d-FFR — Measure FFR and d-FFR

SUMMARY:
This study clarified the influence of myocardial bridge on coronary hemodynamics by clarifying FFR and d-FFR to guide clinical intervention and treatment.

DETAILED DESCRIPTION:
Myocardial bridge is a congenital anatomical abnormality, which is generally considered to be a benign change, but individual can cause angina, myocardial infarction and even sudden death. Previously, it was believed that the degree of myocardial ischemia induced by myocardial bridge was related to factors such as the location, length, and systolic stenosis of the myocardial bridge shown by coronary angiography.However, in recent years, more and more evidence has suggested that there is a high degree of mismatch between anatomical stenosis and its function.Studies have shown that FFR and d-FFR can accurately evaluate the functional significance of stenotic lesions.This study intends to enroll patients who underwent coronary angiography due to chest pain and confirmed the left anterior descending artery (LAD) simple myocardial bridge systolic stenosis ≥30%, and the pressure guide wire was used to measure the FFR and d-FFR of the myocardial bridge lesion under static and dobutamine stress.Analyze the relationship between these functional parameters and the anatomical morphological characteristics of the myocardial bridge and other possible clinical influencing factors, and explore the influence of the morphological characteristics of the myocardial bridge on myocardial hemodynamics，so as to clarify the degree of myocardial bridge shown by angiography may induce obvious myocardial ischemia, which requires clinical intensive intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest pain aged ≥18 years old, regardless of gender;
* Coronary angiography shows a solitary myocardial bridge with systolic diameter stenosis ≥30% in LAD;
* Have the ability to complete an ECG exercise test;
* Sign informed consent and are willing to participate in the intended study.

Exclusion Criteria:

* Patients with acute coronary syndrome;
* Coronary angiography shows that the diameter of atherosclerosis in the non-myocardial bridge area of LAD is ≥30%;
* RCA or LCX has severe fixed stenosis, diameter stenosis ≥70% or FFR<0.75, and no interventional therapy is accepted;
* Hypertrophic obstructive cardiomyopathy or more than moderate heart valve disease;
* Atrial fibrillation or severe slow or rapid arrhythmia;
* Heart failure with NYHA ≥ Grade III;
* Uncontrolled hypertension or systolic blood pressure <100mmHg;
* Asthma or severe chronic obstructive pulmonary disease;
* Severe liver and kidney dysfunction;
* Allergic to contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators enrolled patients with LAD simple myocardial bridge after other interventional treatments for vascular lesions or FFR testing to exclude functionally significant lesions.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Morphological index of myocardial bridge | All indicators were completed within 1 week of coronary angiography.
  The minimum lumen diameter of the target vessel

SECONDARY OUTCOMES:
Exercise electrocardiogram | 72 hours after coronary angiography
  ST segment depression time

CONTACTS AND LOCATIONS:
Overall Officials: Liyun He, Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No